CLINICAL TRIAL: NCT05632627
Title: Cannabinoids and Traumatic Brain Injury: A Randomized, Placebo Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-1427
Record Dates: First submitted 2022-10-24; First posted 2022-11-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Brain Injuries, Traumatic
Keywords: TBI; CBD
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full Spectrum Cannabidiol (Active Comparator): Full Spectrum Cannabidiol (<0.3% THC) Oral softgel capsule, 210mg/day
  Interventions: Drug: Cannabidiol
- Broad Spectrum Cannabidiol (Active Comparator): Broad Spectrum Cannabidiol (0.0% THC) Oral softgel capsule, 210mg/day
  Interventions: Drug: Cannabidiol
- Hemp Seed Oil (Placebo Comparator): Placebo Oral softgel capsule, 210mg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The current study will directly test the hypothesis that a moderate dose of CBD leads to improvements in cognition, TBI-related symptoms, pain, sleep, depression, anxiety, and peripheral markers of inflammation and oxidative stress.
  Other Names: CBD
  Arms: Broad Spectrum Cannabidiol; Full Spectrum Cannabidiol
Drug: Placebo — Placebo arm
  Arms: Hemp Seed Oil

SUMMARY:
This is a double-blind, placebo-controlled, parallel group study designed to assess the tolerability and efficacy of fsCBD and bsCBD, compared to a placebo control, to improve cognition and traumatic brain injury-related symptoms. If eligible for the study, subjects will be randomized to receive one of the conditions for 12 weeks.

DETAILED DESCRIPTION:
To better understand the effects of hemp-derived CBD with and without a small amount of THC, we propose a Phase II randomized clinical trial (RCT) to examine the safety, tolerability, and clinical effects of Full Spectrum CBD (fsCBD, contains less than 0.3% THC) vs. Broad Spectrum CBD (bsCBD, does not contain THC), vs. a matching placebo in a population of patients with traumatic brain injury.

This is a double-blind, placebo-controlled, parallel group study designed to assess the tolerability and efficacy of fsCBD and bsCBD, compared to a placebo control, to improve cognition and TBI-related symptoms such as anxiety, pain, depression, and sleep. If eligible for the study, subjects will be randomized to receive one of the conditions for 12 weeks.

The initial Week 0 / Baseline visit will take place at the University of Colorado Anschutz Medical Campus. There will be in-person visits at Weeks 1, 6, and 12. Participants will be contacted remotely each remaining week during the 12-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide valid informed consent
2. 18-60 years old
3. Current or history of TBI as identified by the Ohio Identification Method
4. TBI severity is mild or moderate based on the VA/DoD Classification of TBI Severity
5. TBI event must have resulted in hospital evaluation (emergency department or other hospital-based assessment) or evaluation within a clinical setting, except in cases in which the TBI was acquired in a military deployment context in which medical services were not immediately available
6. Ongoing neuropsychiatric symptoms (i.e., depressive, anxiety, pain, cognitive complaints, or sleep complaints) that are plausibly associated with TBI and not better accounted for by co-occurring medical or psychological health conditions
7. Not currently in another treatment study for TBI-related symptoms or co-occurring medical or psychological health conditions
8. Co-occurring treatments must be stable in type, dose, and frequency for the four weeks preceding study enrollment and participants must commit to making no changes in these co-occurring treatments during the study

Exclusion Criteria:

1. Currently incarcerated, paroled, or on probation
2. Participant has retained an attorney in relation to the TBI
3. Pregnant at the time of study enrollment or unwilling to commit to the use of two forms of contraception throughout the duration of the study
4. Vision, hearing, or communication impairments that preclude valid completion of study assessments
5. History of autism spectrum disorders, intellectual disability, and/or serious neurological or central nervous system disease that would be expected to affect cognition (e.g., epilepsy, tumors, multiple sclerosis)
6. Evidence of poor effort (TOMMe < 8) on neuropsychological testing at baseline/Week 0
7. Current or lifetime diagnosis of a schizophrenia spectrum disorder, psychotic disorder, bipolar disorder type I & II, cluster B personality disorders (antisocial, borderline, narcissistic, histrionic), eating disorders, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revised (DSM-5-TR, APA 2022)
8. Meets criteria for major depressive episode as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revised (DSM-5-TR, APA 2022) and with a Beck Depression Inventory-2 score > 24;
9. Current suicidal ideation, as indicated by Beck Depression Inventory-2 item #9 score > 0, or C-SSRS endorsement of item #2, or verbal or written report of current suicidal ideation by the participant to any study team member
10. History of significant systemic illness or unstable medical condition
11. Alcohol use disorder score of 5 or greater, or substance use disorder, based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revised (DSM-5-TR, APA 2022), in the six months preceding study enrollment
12. Reported use of other drugs (cocaine, opiates, methamphetamine, MDMA) in the past 60 days or test positive on a urine test for those drugs of abuse at baseline;
13. Currently taking medications known to be contraindicated with Epidiolex (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, teriflunomide, clobazam, lamotrigine, valproate).
14. Current diagnosis of a seizure disorder or epilepsy
15. Report using cannabis once daily or more than once daily over the last 12 months
16. Report current use of CBD for medical reasons or TBI symptoms
17. Liver function enzymes (AST, ALT) that are greater than 2x normal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Neuropsychiatric Symptoms | Week 0 to Week 12
  The effects of study treatment (CBD or placebo) on neuropsychiatric symptoms associated with TBI will be assessed by the Neurobehavioral Symptom Inventory (NSI)
Change in Cognition | Week 0 to Week 12
  The effects of study treatment (CBD or placebo) on attention, processing speed, working memory, long-term memory recall, and executive function will be assessed using the Trail Making Test; the Wechsler Adult Intelligence Scale-IV (WAIS-IV) Digit Span, Symbol Search, Coding, Letter-Number Sequencing; and HVLT delayed recall, to create domain scores used to inform an aggregate measure of cognition.

SECONDARY OUTCOMES:
Change in Biomarkers of Inflammation | Week 0 to Week 6, Week 0 to Week 12
  Circulating levels of cytokine proteins before and after will be measured using immunoassay before and after treatment
Change in Biomarkers of Oxidative Stress | Week 0 to Week 12
  Circulating levels of cytokine proteins before and after will be measured using immunoassay before and after treatment
Change in Pain Intensity | Week 0 to 12
  PROMIS Pain Intensity 1a - A single-item measure of pain intensity. Average pain in the last 7 days is recorded on a scale of 1 - 10, with higher scores indicating higher pain levels.
Change in Anxiety | Week 0 to 12
  PROMIS Anxiety SF - An 8-item measure to rate subjective anxiety symptoms. Possible scores range from 1 - 5 with higher scores indicating worse anxiety symptoms.
Change in Sleep Disturbance | Week 0 to Week 6, Week 0 to Week 12
  PROMIS SF v10 Sleep Disturbance 4a - a 4-item measure assessing subjective sleep quality.
Change in Quality of Life | Week 0 to Week 12
  The Short Form 36 will be used to measure quality of life.
Change in Depression | Week 0 to Week 12
  The Beck Depression Inventory II (BDI-II) will be used to measure depressive symptoms throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hutchison, PhD, Principal Investigator — kent.hutchison@cuanschutz.edu
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No